CLINICAL TRIAL: NCT02724306
Title: A Randomised Controlled Trial Investigating the Effect of a 12 Month Active Lifestyle Programme on Physiological Risk Markers and Physical Activity Behaviour in Those Diagnosed With Intermediate or High Risk for Colon Cancer
Brief Title: Physical Activity Intervention With People at Increased Risk of Developing Colon Cancer
Acronym: PARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12/EE/0106
Record Dates: First submitted 2016-02-12; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Colon Polyps; Colon Adenomas
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Lifestyle Programme (Experimental): ALP will receive supervised exercise sessions twice per week for three months and once per week for the following three months. Participants will also take part in biweekly physical activity workshops for the period of the intervention. Each session consists of a warm-up (5-10min), aerobic (20-30min) and resistance exercises (15-20), and cool-down (5-10)stretches lasting in total 60min. The intensity of exercises will be at 65-85% of maximum heart rate as determined by maximal fitness test. Exercise will take place in small groups of two to five people. Behaviour change workshops to aid the uptake and maintenance of physical activity will be delivered every fortnight throughout the whole intervention period totalling 12 workshops. Workshops will also take place in small groups.
  Interventions: Behavioral: Active Lifestyle Programme
- Standard Care (No Intervention): The standard care group will not be offered the intervention until the end of the study at 12 months. Participants in this group will be encouraged to continue with their usual lifestyle.

INTERVENTIONS:
Behavioral: Active Lifestyle Programme
  Arms: Active Lifestyle Programme

SUMMARY:
The present study will use a randomised controlled trial design to investigate whether moderate to vigorous intensity physical activity (MVPA) will affect the physiological risk markers associated with the development of bowel cancer in individuals previously diagnosed with a bowel polyp. The study will also investigate the effects of the programme on long-term exercise behaviour and changes in psychological variables. A selected sample will also be part of individual interviews at baseline and 12 months to gauge narrative accounts of personal, psychological and sociological beliefs surrounding participation in physical activity. The findings of this study might inform better practices for the prevention of bowel cancer in high risk populations.

After a screening colonoscopy, eligible participants will be randomised to either an active lifestyle programme (ALP) or a standard care group (SC). Participants in ALP will be offered supervised exercise sessions and motivational interviewing for 6 months. Intervention components will cease after 6 months, but participants will be followed-up at 12 months to investigate maintenance to physical activity over the long-term. The SC will not be offered the intervention until the end of the study. Participants in both groups will be invited for assessments at baseline, 3, 6, 9, and 12 months. These include measurements of body composition, cardiopulmonary fitness, physical activity behaviour, and psycho-social variables.

DETAILED DESCRIPTION:
Purpose: A strong body of evidence suggests that lifestyle factors influence cancer risk, and there is now convincing evidence that a physically activity lifestyle is associated with reduced risk of developing colon cancer. However, low self-reported physical activity levels in elderly populations demonstrate the need for physical activity interventions for this patient group that evoke meaningful changes in physical activity behaviour for improvements in CC risk profile to occur.

The purpose of this study is to investigate the effects of a 6 month physical activity intervention on physical activity behaviour and biological markers of CC risk in individuals classified as being at elevated risk of developing the disease following surveillance colonoscopy. The physical activity intervention will be underpinned by Self Determination Theory to create an autonomy-supportive environment, an approach that was recently shown to evoke greater physical activity levels and weight loss than general health education in overweight women. Secondary outcomes will explore the impact of the intervention on aerobic fitness, health-related quality of life and psychological variables (self-efficacy, motivational regulation). In addition, interviews and focus groups will be used to obtain narrative accounts of patient experiences, their perceived health benefits from participating in the intervention and the barriers and facilitators influencing adherence.

Design The proposed study is a randomised controlled trial, with participants stratified for risk status (determined by number and size of polyps identified by colonoscopy). Participants will be randomly allocated to either the physical activity intervention (Active Lifestyle Programme: ALP) or the usual care control group (SC). Outcomes will be assessed at baseline, and after 3, 6, 9 and 12 months. Participants allocated to the ALP group will attend supervised exercise sessions at a facility at the University of East Anglia. These will take place twice per week for 3 months and once per week for an additional 3 months. These will be supplemented by home based exercise to achieve a total of 300 minutes of physical activity each week. Supervised exercise sessions will take place in small groups of maximum 7 participants, and last approximately 60 minutes. The exercise sessions will include a 5-10min warm-up period, followed by 20-30 min aerobic exercise, and 15-20 min resistance exercises. The target intensity of the exercises will be 65-85% of the maximum heart rate as determined by the cardiopulmonary fitness test. Intensity will be monitored with heart rate monitors and the rate of perceived exhaustion (Borg Scale). A short cool-down period will conclude the exercise sessions. In addition, participants will be offered physical activity counselling workshops which will be led in groups, and in a motivational interviewing style. All components of the intervention will be undermined by Self-determination Theory, that is to facilitate feelings of autonomy, competence and relatedness.

To further facilitate behaviour change, participants in the ALP group will be provided with pedometers and an educational workbook, which contains information about the benefits of physical activity in general and in regards to bowel cancer, aids to set personalised goals, and other information relevant to physical activity.

There will also be a purposefully selected sample chosen based on prior consent and demographic variables to take part in face to face interviews at 1 and 12 months. Furthermore 3 focus groups containing, participants from the EX and UC group will take place alongside a focus group with Health professionals after the intervention has taken place.

Recruitment and Consenting Potential participants will either hear about the study via posters and flyers at the Big C Cancer Charity at NNUH or they will be approached by a specialist nurse during a consultation appointment before their colonoscopy. However, the recruitment procedure will be the same for each path from the point of their pre-colonoscopy consultation appointment.On the day of the consultation, a nurse will inform the potential participants about the study and give them an invitation letter, and a participant information sheet. At this meeting, the nurse will also provide the patient with a consent form, asking for their agreement to be contacted by a researcher. If the patient gives consent to be contacted, a researcher will call the patient prior to their screening colonoscopy to provide further information about the study, and arrange an appointment to obtain consent for biopsies to be taken during their colonoscopy. If the patient is diagnosed with polyps during the screening colonoscopy, the researcher will arrange another appointment post-colonoscopy to carry out baseline assessments and obtain full study consent.

Baseline assessments will include a maximal fitness test, assessment of current physical activity using accelerometers and self-report, questionnaires assessing quality of life and psycho-social variables, and body composition.

After the completion of all baseline assessments, participants will be randomised to one of the two study arms. This will be carried out by a person not directly involved in the research. The person undertaking the maximal fitness test will be blinded to group allocation throughout the whole duration of the study. The person carrying out the intervention will not be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of 'intermediate' to 'high' risk as a result of the screening colonoscopy-
* aged 60 years and above
* physically able to partake in regular exercise

Exclusion Criteria:

* assignment into the 'low risk' category or diagnosis of colorectal cancer following the colonoscopy;
* physical activity levels of at least 150min per week for the last 6 months
* presence or history of other co-morbid conditions which might preclude patients from safely undertaking regular exercise, including cardiovascular or pulmonary disease or stroke
* presence of other colorectal conditions (e.g. inflammatory bowel disease) or known familial colorectal cancer syndrome
* chronic use of any treatments or alternative therapies that may affect the results of any study of colorectal tissue e.g. high corticosteroid, anticoagulant or laxative use, regular enemas, high dose vitamin or antioxidant supplements, etc.;
* previous diagnosis of cancer;
* inability to adequately understand written and spoken English,
* presence of drug controlled type II diabetes mellitus
* current involvement in other ongoing research

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in DNA methylation in genes associated with inflammation and colon carcinogenesis | 0, 6, 12 months
Compliance to intervention | post-intervention (at 6months)
  Physical activity diary used to assess compliance
Change in minutes spent in moderate and vigorous intensity physical activity measure with the International Physical Activity Questionnaire long version | 0, 3, 6, 9,12
Change in minutes spent in moderate and vigorous intensity leisure activity assessed with the Godin Leisure-Time Exercise Questionnaire | 0, 3, 6, 9, 12

SECONDARY OUTCOMES:
Change in behavioural regulation measure with the Behavioural Regulation in Exercise Questionnaire version 2 | 0, 3, 6, 9, 12 months
Change in Quality of life measure with the SF-36 questionnaire | 0, 3, 6, 9, 12 months
Changes in anthropometric measures (height, weight, BMI) | 0, 3, 6, 9, 12 months
  Body weight and body height will be used to calculate BMI
Change in physical fitness | 0, 6, 12 months
  Assessed with a maximal cardiopulmonary exercise test on a bicycle ergometer
Change in intention to exercise | 0, 3, 6, 9, 12 months
  Intention to exercise scale
Change in barriers to exercise | 0, 3, 6, 9, 12 months
  Assessed with Barriers to Exercise questionnaire
Change in minutes of physical activity measured with objective measure (accelerometer, Actigraph) | 0, 3, 6, 9, 12 months
Changes in body composition (% body fat) assessed with bioelectrical impedance analysis | 0, 3, 6, 9, 12 months
Change in antropometric measures (waist circumference, hip circumference) | 0, 3, 6, 9, 12 months
  Waist and hip circumference will be used to calculate the waist-to-hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: John M Saxton, PhD, Principal Investigator — University of Northumbria

IPD SHARING:
Plan to Share IPD: No